CLINICAL TRIAL: NCT06752629
Title: Comparison Between Dexmedetomidine and Fentanyl As an Adjuvant to Bupivacaine in the Paravertebral Nerve Block in Laparoscopic Cholecystectomy for Postoperative Analgesia: Randomized Comparative Clinical Trial.
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eithar Mahmoud Abd-Elsalm, resident doctor at Assiut University hospital, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: dexm VS fenta cholecystectomy
Record Dates: First submitted 2024-12-11; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Laparoscopic Cholecystectomy
Keywords: paravertebral nerve block
MeSH Terms: interventions — Bupivacaine; Dexmedetomidine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- group 1 (Experimental): Adult patients will take 10 ml Bupivacaine 0.5% plus 2ml solution of Dexmedetomidine 1mic/kg in the bilateral T5&6 preoperatively
  Interventions: Drug: Bupivacaine and Dexmedetomidine
- group 2 (Experimental): Adult patients will take 10 ml Bupivacaine 0.5% plus 2ml solution of Fentanyl 20 microgram with the bilateral T5&6 preoperatively.
  Interventions: Drug: Bupivacaine and Fentanyl

INTERVENTIONS:
Drug: Bupivacaine and Dexmedetomidine — Adult patients will take 10 ml Bupivacaine 0.5% plus 2ml solution of Dexmedetomidine 1mic/kg in the bilateral T5&6 preoperatively
  Arms: group 1
Drug: Bupivacaine and Fentanyl — Adult patients will take 10 ml Bupivacaine 0.5% plus 2ml solution of Fentanyl 20 microgram with the bilateral T5&6 preoperatively
  Arms: group 2

SUMMARY:
Laparoscopic cholecystectomy is one of the most common surgeries today, cause it has many advantages over open cholecystectomy. Although these advantages pain remains a big problem after laparoscopic cholecystectomy which causes patient admission or readmission. This post-operative laparoscopic cholecystectomy pain causes extreme patient discomfort, extended post-anesthesia care unit stay and restricts early recovery.

To overcome this problem, there were trials of inta abdominal instillation with local anesthetics with no positive results , so they combined this with local infiltration at the laparoscopic access sites with no satisfactory postoperative analgesia.

The aim of this study is to evaluate the effect and the difference between dexmedetomidine and fentanyl in pre-operative unilateral (T5&6) thoracic paravertebral block for postoperative analgesia in laparoscopic cholecystectomy

DETAILED DESCRIPTION:
The para-vertebral block has been largely used over the past years for post-operative analgesia. Many reports in the literature describe the use of thoracic paravertebral block for providing post-laparoscopic cholecystectomy analgesia. Thanks to the ultrasound, over the past years, paravertebral blocks (PVB) have been increasingly used for providing postoperative analgesia, and in the administration of thoracic paravertebral block which has greatly reduced the incidence of associated complications.

Contrary to the intra-abdominal instillation of local anesthetics and local infiltration, the paravertebral blockade has been reported to provide high-quality afferent blockade with the abolishment of somatosensory evoked potentials. and has also been found capable of attenuating the postoperative stress response associated with traditional cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients within age; (18-60)
* Body mass index (BMI); (18-30)
* ASA I - II

Exclusion Criteria:

* ● Patient refusal to participate in the study

  * Allergy to local anesthetics
  * Coagulopathy
  * Morbid obesity
  * Decreased pulmonary reserve
  * Cardiac disorder
  * Renal dysfunction
  * Pre-existing neurological deficit
  * Psychiatric illness

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
level of sensory block duration | 48 hours
  We will evaluate the sensory block by counting the number of dermatomes at regular intervals . Dermatome regression will be used as a marker of sensory block.

IPD SHARING:
Plan to Share IPD: Undecided